CLINICAL TRIAL: NCT00677508
Title: Development of an Instrument to Measure Quality of Life in Children With Chronic Constipation and Soiling
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry); University of South Alabama (Other); Boston Children's Hospital (Other); Ohio State University (Other); University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Manu Sood, Chief, Associate Professor, Medical College of Wisconsin
Other Study IDs: CHW 05/154
Record Dates: First submitted 2008-05-09; First posted 2008-05-14 (Estimated); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Constipation; Fecal Incontinence
Keywords: Constipation; Fecal incontinence; Quality of life; Health related quality of life
MeSH Terms: conditions — Constipation; Fecal Incontinence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- C FR: Children with constipation and fecal incontinence.
- C: Children with constipation but without fecal incontinence.
- P-C FR: Parents of children with constipation and/or fecal incontinence.

SUMMARY:
We propose to develop parent and child disease-specific instruments to assess health related quality of life (HRQoL) in children with constipation and fecal incontinence.

DETAILED DESCRIPTION:
Chronic constipation is a common problem in childhood, accounting for almost 3% of consultations in pediatric practice. In many children constipation is accompanied by overflow soiling (fecal incontinence). This condition often gives rise to behavioral, social, and emotional problems.

We plan to develop a disease-specific instrument to assess HRQoL in children with constipation and fecal incontinence. We hypothesize that HRQoL is worse in children with fecal incontinence compared to children with constipation but no fecal incontinence. The instrument will involve both parent and child self-reporting measures and will enable researchers to evaluate how disease and treatment strategies impact both child and parent perceptions of quality of life. In the long run this will enable physicians to develop a child friendly approach to management of chronic constipation and fecal incontinence.

ELIGIBILITY:
Inclusion criteria:

1. Age 2-18 years
2. Child and parents fluent in English
3. Child must meet one of the following criteria;

A. Constipation and fecal incontinence: must include 2 or more of the following in a child with insufficient criteria for a diagnosis of IBS (criteria fulfilled at least once per week for at least 2 months before diagnosis in a child over 4 years of age and for at least one month in a child less than 4 years of age):

1. Two or fewer defecations in the toilet per week
2. At least 1 episode of fecal incontinence per week
3. History of retentive posturing or excessive volitional stool retention
4. History of painful or hard bowel movements
5. Presence of a large fecal mass in the rectum
6. History of large diameter stools that may obstruct the toilet

B. Constipation predominant IBS: must include the following, once a week for at least 2 months:

1. Abdominal pain/discomfort, associated with 2 of the following:

   * improved with defecation
   * onset associated with 2 or less stools per week
   * onset associated with hard or lump stool
2. no evidence of inflammatory, anatomic, metabolic or neoplastic processes.

C. Non retentive fecal incontinence: must include all of the following in a child with a developmental age of at least 4 years (criteria fulfilled at least once per week for at least 2 months before diagnosis) [4]:

1. Defecation into places inappropriate to the social context at least once per month.
2. No evidence of an inflammatory, anatomic, metabolic, or neoplastic process that explains the subject's symptoms
3. No evidence of fecal retention.

Exclusion criteria:

1. Children with developmental delays and children over 12 years of age who are unable to understand the questionnaires.
2. Associated chronic disease which may have an impact on quality of life such as cerebral palsy, spine deformity or malformations, learning difficulties, severe mental illness, celiac disease, etc.
3. Child and parents not fluent in English.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children will be recruited from the Constipation Clinic at Children's Hospital of Wisconsin, as well as four coolaborating sites.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2005-09 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To develop and validate child and parent questionnaires to assess HRQoL of children with chronic constipation and fecal incontinence. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Manu Sood, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Treurniet HF, Essink-Bot ML, Mackenbach JP, van der Maas PJ. Health-related quality of life: an indicator of quality of care? Qual Life Res. 1997 May;6(4):363-9. doi: 10.1023/a:1018435427116. PMID 9248318
- [Background] Brooks RC, Copen RM, Cox DJ, Morris J, Borowitz S, Sutphen J. Review of the treatment literature for encopresis, functional constipation, and stool-toileting refusal. Ann Behav Med. 2000 Summer;22(3):260-7. doi: 10.1007/BF02895121. PMID 11211851
- [Background] Youssef NN, Langseder AL, Verga BJ, Mones RL, Rosh JR. Chronic childhood constipation is associated with impaired quality of life: a case-controlled study. J Pediatr Gastroenterol Nutr. 2005 Jul;41(1):56-60. doi: 10.1097/01.mpg.0000167500.34236.6a. PMID 15990631